CLINICAL TRIAL: NCT00890461
Title: Reconstruction of 12-Lead Electrogram From Intracardiac Signals From Defibrillators During or After Implantation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Samir Saba, Director, Cardiac Electrophysiology, UPMC, University of Pittsburgh
Other Study IDs: PRO07080211
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: ICD
Keywords: ECG; ICD
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Defibrillator: The subject population will be obtained by approaching the Principal and Co- Investigators' patients who have been referred for ICD implantation or who already have an ICD. This population ranges in age from 18 years on, and includes both males and females. A maximum of 50 subjects will be enrolled in this study.
  Interventions: Radiation: CT scan of the chest without contrast

INTERVENTIONS:
Radiation: CT scan of the chest without contrast — Patients consenting to participate in the study may also undergo a baseline CT scan of the cest without contrast to allow for the geometrical characterization of their intracardiac electrodes from the ICD system in relation to the position of the 12-lead surface ECG electrodes which would be applied to the chest prior to the CT scan. This scan involves a small amount of radiation, a dose of approximately 1 rem. For comparison, radiation workers are permitted, by federal regulation, a maximum annual radiation exposure of 20 rems to the most sensitive organs of their body.
  Other Names: CT scan; ECG; ICD

SUMMARY:
The purpose of this study is to reconstruct a 12-lead electrocardiogram (ECG) from intracardiac (IC) electrograms (EGM) obtained from defibrillator devices (ICD). The purpose of such a reconstruction is to allow the use of IC EGM for diagnosis of clinical conditions for which ECG have historically been used, and to test the feasibility of a reconstruction technique for the standard 12-lead or extended electrocardiogram from electrical potentials obtained from inside a patient.

DETAILED DESCRIPTION:
Reconstructing a 12-lead surface ECG from intracardiac EGM vectors of patients implanted with defibrillators can be of great value. It allows implantable devices that have thus far been used exclusively for arrhythmia detection and treatment, to be used for diagnostic purposes in similar ways as the ECG. The advantage of the reconstruction process is that it provides real-time continuous monitoring, which can be used for multiple purposes, including but not limited to:

1. Ischemia detection
2. Myocardial Infarction detection
3. Electrolyte abnormalities detection
4. Assessment of effect of medications
5. Improved rhythm discrimination

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age.
2. Subjects must be referred for ICD implantation or already have an ICD implanted..
3. Subjects must be willing to sign informed consent.

Exclusion Criteria:

1. Subject is unable or unwilling to sign informed consent.
2. Subject is pacemaker dependent.
3. Subject is pregnant as indicated by standard clinical procedures prior to implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified by their cardiologist who is also an investigator on this study at the time they are evaluated for an ICD implantation. Once it has been determined during the course of the patient's regular clinical care that he or she requires an ICD, they will be approached for enrollment into the study by the physician investigator and the clinical research coordinator.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir F Saba, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania